CLINICAL TRIAL: NCT05354544
Title: A Pilot Study Evaluating the Safety and Feasibility of Autologous Stromal Vascular Fraction in Subjects with Vocal Fold Scar
Brief Title: Evaluating Autologous Stromal Vascular Fraction in Subjects with Vocal Fold Scar
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding loss
Sponsor: Shane A. Shapiro (Other)
Responsible Party: Sponsor-Investigator, Shane A. Shapiro, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-006564
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-06

CONDITIONS: Vocal Fold Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SVF for treating scarred vocal folds (Experimental): Subject identified with scarred vocal folds will have autologous adipose derived SVF harvested and applied to scarred vocal folds.
  Interventions: Biological: Autologous adipose derived SVF

INTERVENTIONS:
Biological: Autologous adipose derived SVF — A single dose of autologous adipose derived SVF isolated from adipose tissue will be administered to scarred vocal folds.

SUMMARY:
The purpose of this research study is to assess if autologous Stromal Vascular Fraction (SVF) taken from the stomach or hips can help heal vocal fold scars.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subject's age between 18 and < 80-years-old
* Voice handicap index greater than 10/40
* Scarred vocal folds or congenital sulcus or after vocal fold surgery (Scarring will be scored during examination and identification of scarred vocal folds and hoarseness. This criterion includes the lack of or decreased mucosal wave of the vocal fold during videostroboscopy exam. Scoring of scar based on laryngoscopic exam: Type I: atrophy of lamina propria with/without affected epithelium. Type II: the epithelium, lamina propria, and muscle are affected. Type III: scar located on the anterior commissure. Type IV: this category includes extended scar formation in both anteroposterior and rostro-caudal axis, with significant loss of vocal fold mass)
* Unilateral or Bilateral vocal fold scarring
* At least 1-year delay after initial surgery
* Negative pregnancy test and contraception for woman of childbearing age. Women of childbearing age must use contraception at least 4 months pre and post SVF administration.

Exclusion Criteria:

* Refusal of speech therapy
* History of malignant lesion or severe dysplasia of the scarred vocal fold
* Contraindication to anesthesia, anticoagulant treatment, coagulation disorders, active infectious disease
* Refusal or inability to comply with study procedures
* Pregnant and lactating woman
* Major chronic medical condition that could affect treatment or quality of SVF product. These include:

  * Current treatment or within 6 months of last treatment for cancer.
  * Blindness
  * Known history of Dementia,
  * Known history of Kidney Disease
  * Known history of Cerebral Vascular Accident or Stroke
* Known history of Diabetes
* Abnormal screening lab. If the laboratory reports a single, non-clinically relevant, non-life-threatening result for any of these studies and is the only excluding factor it may be repeated 1 week later if the subject wishes. Normalization of that laboratory study will then be considered non-exclusionary.
* Post-Radiation scarring of vocal folds.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Adverse events post SVF administration | 24 months
  Number of adverse events related to SVF via endoscopy into vocal folds defined as inflammation or swelling indicated by red or swollen vocal folds or evidence of a hemorrhage indicated by a bleed at or near the site of delivery. This will be evaluated during stroboscope exam.

SECONDARY OUTCOMES:
Voice handicap Index | Baseline, Week 1, and Months 1, 3, 6, 9, 12, and 24
  Change in the self-reported voice handicap index to describe voices and effects of voices on subject lives, measure using a total score range from 0-120; 0-30=mild, 31-60=moderate, 60-120=severe

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rutt, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials